CLINICAL TRIAL: NCT05080582
Title: Does Mother Scented Simulated Hand Promote Comfort, Reduce Pain and Distress Among Mechanically Ventilated Preterm Neonates During Invasive Procedures
Brief Title: Mother Scented Simulated Hand for Mechanically Ventilated Preterm Neonates During Invasive Procedures?
Acronym: Zaky-Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Pediatric nurse specialist, Faculty of Nursing, principal Investigator, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1614032021
Record Dates: First submitted 2021-09-28; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Pain; Distress, Emotional
Keywords: Simulated Hand; Comfort; Pain; Distress; Invasive procedures; Preterm Neonates
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother-Scented Simulated Hand (Experimental): The neonates received the same standard care of the NICU, while they wrapped with a warm Mother-Scented Simulated Hand as follow; simulated hand was scented with mothers' body odor by placing it on the mothers' bare chest or behind the neck for one hour. Then, the MSSH was placed under a radiant warmer for a couple of minutes to reach the mothers' unique warm touch. Inside the incubator, the mechanically ventilated neonates were placed in a side-lying flexed fetal position, where they encircled with the two warm simulated human hand to contain them. Where the palm of one MSSH cupped the neonates' head, and the palm of the other hand cupped the lower part of body and extremities. The neonates were kept in such a position throughout the mentioned invasive procedures, as shown in Figure 2. Neonates' physiological response, comfort, distress, and pain levels were assessed the same way as the first day.
  Interventions: Behavioral: Mother-Scented Simulated Hand
- NICU Standard Care (Active Comparator): The neonates were provided with standard care, which entailed maintaining a quiet environment with minimal stimulation, uninterrupted periods of sleep, containment. Neonates were placed in a side-lying position, while their extremities were flexed close to the body and wrapped with rolled sheets or towels to simulate the intrauterine posture. This position was maintained during the performance of the invasive procedures.
  Interventions: Behavioral: NICU Standard Care

INTERVENTIONS:
Behavioral: Mother-Scented Simulated Hand — Preterm neonates wrapped with a warm Mother-Scented Simulated Hand during the invasive procedures
  Arms: Mother-Scented Simulated Hand
Behavioral: NICU Standard Care — Neonates were placed in a side-lying position, while their extremities were flexed close to the body and wrapped with rolled sheets or towels to simulate the intrauterine posture.
  Arms: NICU Standard Care

SUMMARY:
This study aimed to determine the effect of Mother-Scented Simulated Hand (MSSH) on promoting comfort among mechanically ventilated preterm neonates during invasive procedures.

Research Hypotheses

* Preterm neonates who receive MSSHH exhibit higher levels of comfort during invasive procedures than those who receive standard care.
* Preterm neonates who receive MSSHH exhibit lower levels of pain and stress during invasive procedures than those who receive standard care

DETAILED DESCRIPTION:
A quasi-experimental, pre-posttest, two group, study was carried out in NICU of in Smouha, Alexandria. A sample of 62 mechanically ventilated neonates were randomly assigned to two equal groups; the study group wrapped with a warm MSSH during the invasive procedures while the control group received standard care of NICU. Two observers independently rated the neonates' level of comfort, distress, and pain during Endotracheal Suctioning (ETS) and heel prick using COMFORTneo Scale.

On day one of mechanical ventilation, the neonates received the same standard care of the NICU, while they wrapped with a warm Mother-Scented Simulated Hand as follow; simulated hand was scented with mothers' body odor by placing it on the mothers' bare chest or behind the neck for one hour. Then, the MSSH was placed under a radiant warmer for a couple of minutes to reach the mothers' unique warm touch. Inside the incubator, the mechanically ventilated neonates were placed in a side-lying flexed fetal position, where they encircled with the two warm simulated human hand to contain them. Where the palm of one MSSH cupped the neonates' head, and the palm of the other hand cupped the lower part of body and extremities. The neonates were kept in such a position throughout the mentioned invasive procedures. Neonates' physiological response, comfort, distress, and pain levels were assessed the same way as the first day.

ELIGIBILITY:
Inclusion Criteria:

* Preterm
* Newly admitted
* Hemodynamic stability

Exclusion Criteria:

* Receiving sedatives
* Low APGAR score lower than three at five minutes
* Hypothermia
* Hypoglycemia
* Hyperglycemia
* Intraventricular hemorrhage grade III& IV
* Neonatal seizures

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Level of comfort, pain and distress | immediately after the intervention
  COMFORTneo Scale:
  This scale was developed by Dijk et al. (2009). It is a numerical rating scale to assess neonates' comfort, distress and pain levels. It consists of 6 items, including alertness, calmness/agitation, respiratory response, body movement, facial tension, and muscle tone. The neonates' behavioral response was rated on 5 points numerical rating scale (1-5), and the total score ranged from 6 to 30. The lower score indicates a higher level of comfort and vice versa.
  The COMFORTneo scale has additional two Numerical Rating Scales (NRSs) for pain and distress. These scales are scored after the COMFORTneo score. Both of them range from zero to ten; the Zero score represents no pain or distress, while the ten score represents the worst imaginable pain or distress.

CONTACTS AND LOCATIONS:
Overall Officials: Eman m Taha, professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu TW, Azhibekov T, Seri I. Transitional Hemodynamics in Preterm Neonates: Clinical Relevance. Pediatr Neonatol. 2016 Feb;57(1):7-18. doi: 10.1016/j.pedneo.2015.07.002. Epub 2015 Aug 29. PMID 26482579
- [Background] Holsti L, Grunau RE, Shany E. Assessing pain in preterm infants in the neonatal intensive care unit: moving to a 'brain-oriented' approach. Pain Manag. 2011 Mar 1;1(2):171-179. doi: 10.2217/pmt.10.19. PMID 21874145
- [Background] Loos HM, Reger D, Schaal B. The odour of human milk: Its chemical variability and detection by newborns. Physiol Behav. 2019 Feb 1;199:88-99. doi: 10.1016/j.physbeh.2018.11.008. Epub 2018 Nov 8. PMID 30414885
- [Background] Pineda R, Bender J, Hall B, Shabosky L, Annecca A, Smith J. Parent participation in the neonatal intensive care unit: Predictors and relationships to neurobehavior and developmental outcomes. Early Hum Dev. 2018 Feb;117:32-38. doi: 10.1016/j.earlhumdev.2017.12.008. Epub 2017 Dec 21. PMID 29275070
- [Background] Zeraati H, Nasimi F, Rezaeian A, Shahinfar J, Ghorban Zade M. Effect of Multi-sensory Stimulation on Neuromuscular Development of Premature Infants: A Randomized Clinical Trial. Iran J Child Neurol. 2018 Summer;12(3):32-39. PMID 30026767
- [Background] Vittner D, Butler S, Smith K, Makris N, Brownell E, Samra H, McGrath J. Parent Engagement Correlates With Parent and Preterm Infant Oxytocin Release During Skin-to-Skin Contact. Adv Neonatal Care. 2019 Feb;19(1):73-79. doi: 10.1097/ANC.0000000000000558. PMID 30335622
- [Background] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803